CLINICAL TRIAL: NCT04015869
Title: Effect of Allopregnanolone on Stress-induced Craving
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Ralevski, Research Scientist, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2000021601; 1R21AA024917-01A1 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-07-11 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Pregnanolone

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- allopregnanolone (Active Comparator): Allopregnanolone infusion dose of 100nM over 175 min
  Interventions: Drug: Allopregnanolone
- placebo (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Allopregnanolone — neurosteroid
  Arms: allopregnanolone
Drug: Placebos — placebo
  Arms: placebo

SUMMARY:
The goal of this study is to determine whether intravenous infusion of allopregnanolone (ALLO) attenuates stress-induced craving and stress-induced anxiety in a clinical laboratory setting. The secondary objective of this project is to characterize the behavioral effects of ALLO in heavy drinkers.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study that will randomize heavy "at risk" drinkers to 2 groups: targeted dose of 100 nM of ALLO or placebo. Participants will receive a continuous infusion of ALLO (or placebo) for approximately 175 min. Sixty minutes after the start of the infusion, when ALLO levels are relatively stable, the stress induction paradigm will be introduced. Participants will be presented with a stress cue and a neutral cue in random order. Stress and neutral cues will consist of personalized 5-minute scripts created prior to testing. Measures of stress-induced craving and stress-induced anxiety will be presented before the cue (pre), immediately following the cue (post) and 10 minutes after (recovery). An alcohol infusion (40mg%) begins at approximately 120 minutes into ALLO Infusion. Once the alcohol infusion has reached the targeted dose of 40mg% the infusion is clamped for approximately 20 minutes. The study outcomes will include measures of stress-induced craving and stress-induced anxiety as well as measures of subjective mood effects, cognitive performance, and motor coordination.

ELIGIBILITY:
Inclusion Criteria:

* Non-treatment seeking individuals with current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) alcohol use disorder (AUD)
* No current substance use disorder (except tobacco, alcohol, and marijuana)
* No current medical problems and normal electrocardiogram (ECG)
* For women, not pregnant as determined by pregnancy screening, not breast feeding.

Exclusion Criteria:

* Current major psychiatric illnesses including mood, psychotic, or anxiety disorders
* History of major medical illnesses; including liver diseases, heart disease, chronic pain or other medical conditions that the physician investigator deems contraindicated for the subject to be in the study
* Liver function tests (ALT or AST) greater than 3 times normal
* weight >120kg
* renal impairment
* patients on the following medications: a) medications for alcoholism (e.g. naltrexone, disulfiram, topiramate, acamprosate); b) psychotropic medications that promote sedation (please note patients on psychotropic medications for current psychiatric conditions will also be excluded); and c) patients currently taking antibiotics or antifungals

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, PhD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healtcase System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Allopregnanolone: On the test day the participant received an allopregnanolone (ALLO) infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
- Placebo: On the test day the participant received a placebo (for allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
Period: Overall Study
Arm/Group | Allopregnanolone | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Allopregnanolone 100nM: Targeted dose of 100 nM of ALLO, a continuous infusion of ALLO for approximately 175 min. Sixty minutes after the start of the infusion, when ALLO levels are relatively stable, the stress induction paradigm will be introduced. Stress and neutral cues will consist of personalized 5-minute scripts created prior to testing. Measures of stress-induced craving and stress-induced anxiety will be presented before the cue (pre), immediately following the cue (post) and 10 minutes after (recovery). An alcohol infusion (40mg%) begins at approximately 120 minutes into ALLO Infusion. Once the alcohol infusion has reached the targeted dose of 40mg% the infusion is clamped for approximately 20 minutes. After 20-minute clamp both infusions will end.
- Placebo: Placebo dose, a continuous infusion of placebo for approximately 175 min. Sixty minutes after the start of the infusion, when ALLO levels are relatively stable, the stress induction paradigm will be introduced. Stress and neutral cues will consist of personalized 5-minute scripts created prior to testing. Measures of stress-induced craving and stress-induced anxiety will be presented before the cue (pre), immediately following the cue (post) and 10 minutes after (recovery). An alcohol infusion (40mg%) begins at approximately 120 minutes into ALLO Infusion. Once the alcohol infusion has reached the targeted dose of 40mg% the infusion is clamped for approximately 20 minutes. After 20-minute clamp both infusions will end.
- Total: Total of all reporting groups
Arm/Group | Allopregnanolone 100nM | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.8) | 40.8 (7.3) | 38.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Urge Questionnaire (AUQ) Pre-script
Description: The Alcohol Urge Questionnaire (AUQ) is an 8-question, self-administered measure of drinking urges. Questions are in the form of a 7-point scale with participants endorsing the extent to which they agree or disagree with statements relating to desire to drink (4 items), expectation of a desired outcome from drinking (2 items), and inability to avoid drinking if alcohol was available (2 items). Total scores range from 8 (strongly disagree) to 56 (strongly agree).
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Allopregnanolone Trauma Script; Placebo Trauma Script: On the test day the participant received an allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
- Allopregnanolone Neutral Script; Placebo Neutral Script: On the test day the participant received a placebo (for allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 24.45 (6.18) | 21.51 (5.05) | 19.15 (6.18) | 26.29 (5.05)

2. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Upset - Pre-Script
Description: The State Trait Anxiety Inventory (STAI-6) is a 6-item self-rated instrument used to assess anxiety state. The STAI-6 questions included: 1. "I feel calm"; 2. "I am tense"; 3. "I feel upset"; 4. "I am relaxed"; 5. "I feel content"; 6. "I am worried". Each of these questions were rated as: a) "not at all"; b) "somewhat"; c) "moderately"; d) "very much". For questions 2, 3, and 6, the scoring was a = 1, b = 2, c = 3, and d = 4.
  For the other 3 questions, the scoring was a = 4, b = 3, c = 2, and d = 1. This outcome is for 3. "I feel upset" (scored individually): the scoring for "I feel upset is: a = 1, b = 2, c = 3, and d = 4 (1 not at all upset to 4 very much upset)
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Allopregnanolone Neutral Script: On the test day the participant received an allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
- Placebo Trauma Script; Placebo Neutral Script: On the test day the participant received a placebo (for allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.4 (0.26) | 1.0 (0.26) | 1.0 (0.26) | 1.4 (0.26)

3. Primary Outcome: Alcohol Urge Questionnaire (AUQ) Post-Script
Description: as for outcome 1
Time Frame: Post-Script 5 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 27.09 (6.10) | 21.50 (7.61) | 14.12 (6.63) | 24.70 (7.61)

4. Primary Outcome: Alcohol Urge Questionnaire (AUQ) Recovery
Description: as for outcome 1
Time Frame: Recovery 10 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 25.65 (6.56) | 25.76 (6.90) | 17.03 (7.14) | 24.70 (7.61)

5. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Sedation Items - Pre-Script
Description: Biphasic Alcohol Effects Scale (BAES) Sedation items - sum of subjective responses - 0(not at all) to 10 (extremely) for 7 sedation related questions regarding effects of alcohol. Total BAES sedation subscale score: 0 (lower sedation) -70 (higher sedation) with higher numbers indicating greater sedative effects of alcohol.
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: Analysis Population Description: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Allopregnanolone: On the test day the participant received an allopregnanolone infusion over 175 minutes. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant). An alcohol infusion (40mg%) begins at approximately 120 minutes into the ALLO infusion. Once target alcohol dose is reached the alcohol infusion will be clamped and continue for approximately 20 mins.
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 6.4 (2.71) | 6.2 (2.71)

6. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Sedation Items
Description: Biphasic Alcohol Effects Scale (BAES) Sedation items - sum of subjective responses - 0(not at all) to 10 (extremely) for 7 sedation related questions regarding effects of alcohol. Total BAES sedation subscale score: 0 (lower sedation) -70 (higher sedation) with higher numbers indicating greater sedative effects of alcohol. Data presented here is mean at 90 minutes.
Time Frame: Pre-infusion (at 0 minutes), during infusion (approximately 20 minutes) and post-infusion (approximately 90 minutes)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 10.6 (3.38) | 5.2 (3.38)

7. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Sedation Items - Target Alcohol Dose (40mg%)
Description: as for outcome 5
Time Frame: Target Alcohol dose (40mg%) 90 minutes after trauma/neutral script is presented
Population: Analysis Population Description: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 5.8 (3.72) | 4.2 (3.72)

8. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Sedation Items - End of Test Day
Description: as for outcome 5
Time Frame: End of test day 150 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 2.8 (2.54) | 6.4 (2.54)

9. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Stimulation Items - Pre-Script
Description: Biphasic Alcohol Effects Scale (BAES) Simulation items - sum of subjective responses - 0 (not at all) to 10 (extremely) for 7 sedation related questions regarding effects of alcohol. Total BAES stimulation subscale score: 0 (lower sedation) -70 (higher sedation) with higher numbers indicating greater stimulating effects of alcohol.
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: Analysis Population Description: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 25.8 (6.8) | 14.2 (6.8)

10. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Stimulation Items
Description: Biphasic Alcohol Effects Scale (BAES) Simulation items - sum of subjective responses - 0 (not at all) to 10 (extremely) for 7 sedation related questions regarding effects of alcohol. Total BAES stimulation subscale score: 0 (lower sedation) -70 (higher sedation) with higher numbers indicating greater stimulating effects of alcohol. Data presented here is mean at 90 minutes.
Time Frame: Pre-infusion (at 0 minutes), during infusion (approximately 20 minutes) and post-infusion (approximately 90 minutes)
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 17.4 (8.18) | 15.6 (8.18)

11. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Stimulation Items - Target Alcohol Dose (40mg%)
Description: as for outcome 9
Time Frame: Target Alcohol Dose (40mg%) 90 minutes after trauma/neutral script is presented
Population: Analysis Population Description: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 26.2 (5.36) | 31.4 (5.36)

12. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Stimulation Items - End of Test Day
Description: as for outcome 9
Time Frame: End of Test Day 150 minutes after trauma/neutral script is presented
Population: Analysis Population Description: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 17.6 (4.18) | 17.4 (4.18)

13. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Upset - Post-Script
Description: as for outcome 2
Time Frame: Post-Script 5 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.6 (0.26) | 1.0 (0.26) | 1.6 (0.26) | 1.4 (0.26)

14. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Upset - Recovery
Description: as for outcome 2
Time Frame: Recovery 10 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.0 (0.26) | 1.0 (0.26) | 1.4 (0.26) | 1.2 (0.26)

15. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Content - Pre-Script
Description: The State Trait Anxiety Inventory (STAI-6) is a 6-item self-rated instrument used to assess anxiety state. The STAI-6 questions included: 1. "I feel calm"; 2. "I am tense"; 3. "I feel upset"; 4. "I am relaxed"; 5. "I feel content"; 6. "I am worried". Each of these questions were rated as: a) "not at all"; b) "somewhat"; c) "moderately"; d) "very much". For questions 2, 3, and 6, the scoring was a = 1, b = 2, c = 3, and d = 4.
  For the other 3 questions, the scoring was a = 4, b = 3, c = 2, and d = 1. This outcome is for 5. "I feel content" (scored individually): the scoring for "I feel content is: a = 4, b = 3, c = 2, and d = 1 (4 not at all content to 1 very much content)
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 3.16 (0.41) | 3.6 (0.39) | 3.0 (0.39) | 2.2 (0.39)

16. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Content - Post-Script
Description: as for outcome 15
Time Frame: Post-Script 5 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 2.2 (0.39) | 3.6 (0.39) | 2.8 (0.39) | 2.8 (0.39)

17. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I Feel Content - Recovery
Description: as for outcome 15
Time Frame: Recovery10 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 3.2 (0.39) | 3.4 (0.39) | 2.4 (0.39) | 2.2 (0.39)

18. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I am Worried - Pre-Script
Description: The State Trait Anxiety Inventory (STAI-6) is a 6-item self-rated instrument used to assess anxiety state. The STAI-6 questions included: 1. "I feel calm"; 2. "I am tense"; 3. "I feel upset"; 4. "I am relaxed"; 5. "I feel content"; 6. "I am worried". Each of these questions were rated as: a) "not at all"; b) "somewhat"; c) "moderately"; d) "very much". For questions 2, 3, and 6, the scoring was a = 1, b = 2, c = 3, and d = 4. For the other 3 questions, the scoring was a = 4, b = 3, c = 2, and d = 1.
  This outcome is for 6. "I am worried" (scored individually): the scoring for "I feel content is: a = 1, b = 2, c = 3, and d = 4 (1 not at all worried to 4 very much worried)
Time Frame: Pre-Script 40 minutes before trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.0 (0.23) | 1.0 (0.23) | 1.2 (0.23) | 1.6 (0.23)

19. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I am Worried - Post-Script
Description: as for outcome 18
Time Frame: Post-Script 5 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.6 (0.23) | 1.0 (0.23) | 1.4 (0.23) | 1.4 (0.23)

20. Primary Outcome: The State-Trait Anxiety Inventory (STAI-6) I am Worried - Recovery
Description: as for outcome 18
Time Frame: Recovery 10 minutes after trauma/neutral script is presented
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopregnanolone Trauma Script | Allopregnanolone Neutral Script | Placebo Trauma Script | Placebo Neutral Script
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | 1.0 (0.23) | 1.0 (0.23) | 1.2 (0.23) | 1.2 (0.23)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Allopregnanolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT04015869/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT04015869/ICF_000.pdf